CLINICAL TRIAL: NCT05291026
Title: Evaluation of mHealth Intervention to Improve Medication Adherence in Type 2 Diabetes in Nigeria: a Randomized Controlled Trial
Brief Title: Mobile Health Intervention for Improved Adherence in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Obafemi Awolowo University (Other)
Responsible Party: Principal Investigator, Madu Ihekoronye, Lecturer, Obafemi Awolowo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: mH22000
Record Dates: First submitted 2022-03-14; First posted 2022-03-22 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Mellitus
Keywords: mobile health; type 2 diabetes; adherence; health education; follow-up
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Health Education

STUDY DESIGN:
Intervention Model Description: All newly-diagnosed type 2 diabetes patients within the one month period following the retrospective document review, were enrolled, provided they gave their informed consent. Study participants were randomly assigned to either of two equal-sized control and intervention cohorts. The Randomizer App software was used to assign participants to the control and intervention groups. The control group received standard of care only. The intervention group received the standard of care in addition to the mobile phone-based health education and follow-up messaging at the frequency of once daily for 6 months.
Who Masked: Participant, Care Provider
Masking Description: Participants knew neither the identity nor the group placement of other participants. The clinicians who provided care for the participants did not know the identity or the group placement of the participants. Investigators/ Outcome assessors were not among the care givers and did not interface physically with either caregivers or study participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Type 2 diabetes patients, 18 years old and above, enrolled in the out-patient, diabetes clinic of the tertiary health facility, receiving only standard of care, and who gave their informed consent
- intervention group (Experimental): type 2 diabetes patients, 18 years old and above, enrolled in the out-patient diabetes clinic of the tertiary health facility, receiving standard of care in addition to a mobile phone - based health education and follow-up messaging on a frequency of once a day corresponding to how often they are expected to take their medications (that is every day), and who gave their informed consent.
  Interventions: Other: mobile phone-based health information

INTERVENTIONS:
Other: mobile phone-based health information — health education and follow-up messaging, randomly assigned to each participant in the intervention arm using a randomization software, delivered once daily, as short message service (sms)
  Other Names: health education, follow-up messaging
  Arms: intervention group

SUMMARY:
The study assessed patients' glycemic control, knowledge of type 2 diabetes (T2D) and adherence to medications, and evaluated the impact of a mobile telephone-based intervention on these indices. Patients' clinic attendance and pharmacy refill records were reviewed for the period of 1 year. Then over a period of 1 month, newly diagnosed T2D patients were enrolled in the prospective phase of the study and randomized into control and intervention groups. A mobile phone-based health education and follow-up package was applied to the intervention group alone for a period of 6 months. Afterwards, both groups were assessed and compared on the study outcome parameters. Same questionnaires were used pre- and post-intervention for primary data collection. Descriptive and inferential statistics were used for data analysis.

DETAILED DESCRIPTION:
Objectives of the Study: The study assessed patients' glycemic control, knowledge of type 2 diabetes (T2D) and adherence to medications, and evaluated the impact of a mobile telephone-based intervention on these indices.

Study design: Randomized controlled trial Study Setting: Diabetes Clinic, Endocrinology Unit, Department of Internal Medicine, Obafemi Awolowo University Teaching Hospital Ile Ife, Osun State Nigeria The study was structured in five stages. Study Duration: Seven months Stage 1: Baseline data Task 1: Baseline data for patients' glycemic control were obtained from one-year retrospective review of 1392 patients' files for glycated haemoglobin (HbA1c) measurements.

Task 2: Patients' baseline adherence data were obtained from one-year retrospective review of pharmacy refill records (clinic attendance) Task 3: Development and validation of research instruments (Questionnaires, Short Message Services (SMS).

Task 4: Recruitment and training of research assistants (2 hours daily for 3 days) Stage 2: Recruitment and randomization of participants Task 1: Enrolment of all newly-diagnosed patients (n = 120), enrolled in the Diabetes Clinic in the period of one month following Stage 1 Task 2: Obtaining of informed consent from all newly-diagnosed patients enrolled in the Diabetes Clinic in the one month following Stage 1 Task 3: Collection of participants' baseline knowledge data using structured questionnaire Task 4: Collection of baseline self-reported adherence data using the adapted 8-point Morisky Medication Adherence Scale (MMAS-8) instrument Task 5: Randomization of consenting participants into two equal (n = 60) control and intervention groups using a randomization software Stage 3: Intervention Task 1: Activation of short message services to participants in the intervention cohort at a frequency of one message per day for the period of 6 months.

Task 2: Follow up on clinic attendances of all participants for the period of 6 months Stage 4: Post-Intervention Review Task 1: Repeat administration of same questionnaires originally administered at Stage 2 to all participants Task 1: Review of participants' clinic attendance and pharmacy refill records Task 2: Review of participants HbA1c measurements from their records Stage 5: Data analysis Task 1: Demographic variables of participants were analyzed using descriptive statistics including frequency and percentages Task 2: Weighted mean scores were used to analyze knowledge and adherence scores Task 3: Two-sample t-test was used to compare pre- and post-intervention scores of knowledge and adherence Task 4: Chi square test was conducted to analyze associations between demographic variables and self-reported adherence data Task 5: Statistical package for the social sciences (SPSS) version 21 for windows software was used for data analysis at the p < 0.05 level of significance

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed of type 2 diabetes for the first time in the month following baseline study
* Male or female, 18 yeas of age and above
* Enrolled in the Out-patient Diabetes Clinic of the Teaching Hospital
* Gave informed consent to participate.

Exclusion Criteria:

* Diagnosed of other disease conditions outside type 2 diabetes
* Below 18 years of age
* Not enrolled in the Out-patient Diabetes Clinic of the Teaching Hospital
* Did not give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure | 6 Months
  Reduction in glycated hemoglobin (HbA1c), measured using blood tests, expressed in mmol/mol (%)

SECONDARY OUTCOMES:
Secondary outcome measure I | 6 months
  Knowledge of diabetes, measured as by the mean score of participants in a questionnaire-based survey
Secondary outcome measure II | 6 months
  Adherence to medication, measured by the mean score of participants in a questionnaire-based survey

CONTACTS AND LOCATIONS:
Overall Officials: Kanayo Osemene, Ph.D., Study Director — Department of Clinical Pharmacy and Pharmacy Administration, Obafemi Awolowo University, Ile Ife Nigeria
Locations (1):
- Obafemi Awolowo University Teaching Hospital Complex, Ile-Ife, Osun State, Nigeria

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

REFERENCES:
- [Background] Inzucchi SE, Bergenstal RM, Buse JB, Diamant M, Ferrannini E, Nauck M, Peters AL, Tsapas A, Wender R, Matthews DR. Management of hyperglycaemia in type 2 diabetes: a patient-centered approach. Position statement of the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetologia. 2012 Jun;55(6):1577-96. doi: 10.1007/s00125-012-2534-0. Epub 2012 Apr 20. No abstract available. PMID 22526604
- [Background] Kharroubi AT, Darwish HM. Diabetes mellitus: The epidemic of the century. World J Diabetes. 2015 Jun 25;6(6):850-67. doi: 10.4239/wjd.v6.i6.850. PMID 26131326
- [Background] Olawuyi AT, Adeoye IA. The prevalence and associated factors of non-communicable disease risk factors among civil servants in Ibadan, Nigeria. PLoS One. 2018 Sep 13;13(9):e0203587. doi: 10.1371/journal.pone.0203587. eCollection 2018. PMID 30212508
- [Background] World Health Organization. Diabetes [Internet]. World Health Organisation, Geneva Switzerland; 2018. Available from: https://www.who.int/news-room/factsheets/ detail/diabetes
- [Background] World Health Organisation. World malaria report 2015. World Health Organisation, Geneva Switzerland; 2016.
- [Background] Asche C, LaFleur J, Conner C. A review of diabetes treatment adherence and the association with clinical and economic outcomes. Clin Ther. 2011 Jan;33(1):74-109. doi: 10.1016/j.clinthera.2011.01.019. PMID 21397776
- [Background] Harande Y. Exploring the Literature of Diabetes in Nigeria: A Bibliometrics Study. African Journal of Diabetes Medicine. 2011; 2:1-4.
- [Background] Mouhtadi BB, Alame MM, Malaeb B, Hallit S, Salameh P, Malaeb D. Physician-community pharmacist collaborative care in diabetes management: a pilot study. J Drug Assess. 2018 Oct 23;7(1):61-65. doi: 10.1080/21556660.2018.1535437. eCollection 2018. PMID 30370175
- [Background] Marciano L, Camerini AL, Schulz PJ. The Role of Health Literacy in Diabetes Knowledge, Self-Care, and Glycemic Control: a Meta-analysis. J Gen Intern Med. 2019 Jun;34(6):1007-1017. doi: 10.1007/s11606-019-04832-y. Epub 2019 Mar 15. PMID 30877457
- [Background] Caruso R, Magon A, Baroni I, Dellafiore F, Arrigoni C, Pittella F, Ausili D. Health literacy in type 2 diabetes patients: a systematic review of systematic reviews. Acta Diabetol. 2018 Jan;55(1):1-12. doi: 10.1007/s00592-017-1071-1. Epub 2017 Nov 11. PMID 29129000
- [Background] Ramaj A, Kamberi F, Behrens J. Effects of Diabetes Education on Emotional Distress in Patients with Type 2 Diabetes-An Experimental Study. Open Journal of Endocrine and Metabolic Diseases. 2019 Feb 19; 9(2):9-20.
- [Background] Hong JS, Kang HC. Relationship between oral antihyperglycemic medication adherence and hospitalization, mortality, and healthcare costs in adult ambulatory care patients with type 2 diabetes in South Korea. Med Care. 2011 Apr;49(4):378-84. doi: 10.1097/MLR.0b013e31820292d1. PMID 21368684
- [Background] Hansen RA, Farley JF, Droege M, Maciejewski ML. A retrospective cohort study of economic outcomes and adherence to monotherapy with metformin, pioglitazone, or a sulfonylurea among patients with type 2 diabetes mellitus in the United States from 2003 to 2005. Clin Ther. 2010 Jul;32(7):1308-19. doi: 10.1016/j.clinthera.2010.07.011. PMID 20678679
- [Background] Juarez DT, Tan C, Davis J, Mau M. Factors Affecting Sustained Medication Adherence and Its Impact on Health Care Utilization in Patients with Diabetes. J Pharm Health Serv Res. 2013 Jun;4(2):89-94. doi: 10.1111/jphs.12016. PMID 23717343
- [Background] Garcia-Perez LE, Alvarez M, Dilla T, Gil-Guillen V, Orozco-Beltran D. Adherence to therapies in patients with type 2 diabetes. Diabetes Ther. 2013 Dec;4(2):175-94. doi: 10.1007/s13300-013-0034-y. Epub 2013 Aug 30. PMID 23990497
- [Background] Fasanmade OA, Dagogo-Jack S. Diabetes Care in Nigeria. Ann Glob Health. 2015 Nov-Dec;81(6):821-9. doi: 10.1016/j.aogh.2015.12.012. PMID 27108149
- [Background] Qiao Y, Steve Tsang CC, Hohmeier KC, Dougherty S, Hines L, Chiyaka ET, Wang J. Association Between Medication Adherence and Healthcare Costs Among Patients Receiving the Low-Income Subsidy. Value Health. 2020 Sep;23(9):1210-1217. doi: 10.1016/j.jval.2020.06.005. Epub 2020 Aug 5. PMID 32940239
- [Background] World Health Organization. Long Term-Therapies: Evidence for Action [Internet]. World Health Organisation, Geneva Switzerland; 2003. Available from: ISBN 92-4-154599-2
- [Background] Lam WY, Fresco P. Medication Adherence Measures: An Overview. Biomed Res Int. 2015;2015:217047. doi: 10.1155/2015/217047. Epub 2015 Oct 11. PMID 26539470
- [Background] Kirkman MS, Rowan-Martin MT, Levin R, Fonseca VA, Schmittdiel JA, Herman WH, Aubert RE. Determinants of adherence to diabetes medications: findings from a large pharmacy claims database. Diabetes Care. 2015 Apr;38(4):604-9. doi: 10.2337/dc14-2098. Epub 2015 Jan 8. PMID 25573883
- [Background] Xu L, Li Y, Dai Y, Peng J. Natural products for the treatment of type 2 diabetes mellitus: Pharmacology and mechanisms. Pharmacol Res. 2018 Apr;130:451-465. doi: 10.1016/j.phrs.2018.01.015. Epub 2018 Feb 13. PMID 29395440
- [Background] Williams JL, Walker RJ, Smalls BL, Campbell JA, Egede LE. Effective interventions to improve medication adherence in Type 2 diabetes: a systematic review. Diabetes Manag (Lond). 2014 Jan 1;4(1):29-48. doi: 10.2217/dmt.13.62. PMID 25214893
- [Background] Anghel LA, Farcas AM, Oprean RN. An overview of the common methods used to measure treatment adherence. Med Pharm Rep. 2019 Apr;92(2):117-122. doi: 10.15386/mpr-1201. Epub 2019 Apr 25. PMID 31086837
- [Background] Walker RJ, Smalls BL, Bonilha HS, Campbell JA, Egede LE. Behavioral interventions to improve glycemic control in African Americans with type 2 diabetes: a systematic review. Ethn Dis. 2013 Autumn;23(4):401-8. PMID 24392600
- [Background] Ni Z, Liu C, Wu B, Yang Q, Douglas C, Shaw RJ. An mHealth intervention to improve medication adherence among patients with coronary heart disease in China: Development of an intervention. Int J Nurs Sci. 2018 Sep 8;5(4):322-330. doi: 10.1016/j.ijnss.2018.09.003. eCollection 2018 Oct 10. PMID 31406843
- [Background] Free C, Phillips G, Felix L, Galli L, Patel V, Edwards P. The effectiveness of M-health technologies for improving health and health services: a systematic review protocol. BMC Res Notes. 2010 Oct 6;3:250. doi: 10.1186/1756-0500-3-250. PMID 20925916
- [Background] Mehas N, Hudmon KS, Jaynes H, Klink S, Downey L, Zillich AJ. Impact of Electronic Medication Reminder Caps on Patient Adherence and Blood Pressure. J Pharm Technol. 2021 Oct;37(5):234-243. doi: 10.1177/87551225211018708. Epub 2021 Jul 31. PMID 34752573
- [Background] NB of S (NBS). Nigeria GDP data, Q1, Q2 2021 [Internet]. 17. National Bureau of Statistics (NBS). 2021 [cited 2022 Jan 10]. Available from: https://nigerianstat.gov.ng/elibrary
- [Background] Islam SM, Lechner A, Ferrari U, Froeschl G, Alam DS, Holle R, Seissler J, Niessen LW. Mobile phone intervention for increasing adherence to treatment for type 2 diabetes in an urban area of Bangladesh: protocol for a randomized controlled trial. BMC Health Serv Res. 2014 Nov 26;14:586. doi: 10.1186/s12913-014-0586-1. PMID 25424425
- [Background] Davis F, Davis F. Perceived Usefulness, Perceived Ease of Use, and User Acceptance of Information Technology. MIS Quarterly. 1989 Sep 1; 13:319.
- [Background] Sangeda RZ, Mosha F, Prosperi M, Aboud S, Vercauteren J, Camacho RJ, Lyamuya EF, Van Wijngaerden E, Vandamme AM. Pharmacy refill adherence outperforms self-reported methods in predicting HIV therapy outcome in resource-limited settings. BMC Public Health. 2014 Oct 4;14:1035. doi: 10.1186/1471-2458-14-1035. PMID 25280535
- [Background] de Oliveira-Filho AD, Morisky DE, Neves SJ, Costa FA, de Lyra DP Jr. The 8-item Morisky Medication Adherence Scale: validation of a Brazilian-Portuguese version in hypertensive adults. Res Social Adm Pharm. 2014 May-Jun;10(3):554-61. doi: 10.1016/j.sapharm.2013.10.006. Epub 2013 Oct 26. PMID 24268603
- [Background] Taber KS. The Use of Cronbach's Alpha When Developing and Reporting Research Instruments in Science Education. Res Sci Educ. 2018 Dec 1; 48(6):1273-96
- [Background] Erdoğan Ö, Araman A. Health beliefs and functional health literacy; Interaction with the pharmaceutical services. Istanbul Journal of Pharmacy. 2017 Oct 18; 47:68-71.
- [Background] Uloko AE, Musa BM, Ramalan MA, Gezawa ID, Puepet FH, Uloko AT, Borodo MM, Sada KB. Prevalence and Risk Factors for Diabetes Mellitus in Nigeria: A Systematic Review and Meta-Analysis. Diabetes Ther. 2018 Jun;9(3):1307-1316. doi: 10.1007/s13300-018-0441-1. Epub 2018 May 14. PMID 29761289
- [Background] Taberna M, Gil Moncayo F, Jane-Salas E, Antonio M, Arribas L, Vilajosana E, Peralvez Torres E, Mesia R. The Multidisciplinary Team (MDT) Approach and Quality of Care. Front Oncol. 2020 Mar 20;10:85. doi: 10.3389/fonc.2020.00085. eCollection 2020. PMID 32266126
- [Background] Centers for Disease Control (CDC). National Diabetes Statistics Report 2020. Estimates of diabetes and its burden in the United States. [Internet]. Centers for Disease Control (CDC); 2020 [cited 2022 Jan 10]. Available from: https://www.cdc.gov/diabetes/pdfs/data/statistics/national-diabetes-statistics-report.pdf
- [Background] Ekpenyong C, Akpan U, Ibu J, Nyebuk D. Gender and age specific prevalence and associated risk factors of type 2 diabetes mellitus in Uyo metropolis, South Eastern Nigeria. DiabetologiaCroatica [Internet]. 2012;41(1). Available from: http://www.sciepub.com/reference/340492
- [Background] Boruett P, Kagai D, Njogo S, Nguhiu P, Awuor C, Gitau L, Chalker J, Ross-Degnan D, Wahlstrom R, Tomson G; INRUD -IAA. Facility-level intervention to improve attendance and adherence among patients on anti-retroviral treatment in Kenya--a quasi-experimental study using time series analysis. BMC Health Serv Res. 2013 Jul 1;13:242. doi: 10.1186/1472-6963-13-242. PMID 23816278
- [Background] Ajisegiri WS, Abimbola S, Tesema AG, Odusanya OO, Ojji DB, Peiris D, Joshi R. Aligning policymaking in decentralized health systems: Evaluation of strategies to prevent and control non-communicable diseases in Nigeria. PLOS Glob Public Health. 2021 Nov 10;1(11):e0000050. doi: 10.1371/journal.pgph.0000050. eCollection 2021. PMID 36962096
- [Background] Chawla SPS, Kaur S, Bharti A, Garg R, Kaur M, Soin D, Ghosh A, Pal R. Impact of health education on knowledge, attitude, practices and glycemic control in type 2 diabetes mellitus. J Family Med Prim Care. 2019 Jan;8(1):261-268. doi: 10.4103/jfmpc.jfmpc_228_18. PMID 30911517
- [Background] International Diabetes Federation. IDF. Clinical practice recommendations for managing type 2 diabetes in primary care. [Internet]. [Cited 2021 Oct 19]. Available from: https://www.idf.org/e-library/guidelines/128-idf-clinical-practice-recommendations-formanaging- type-2-diabetes-in-primary-care.html.
- [Background] Houle SK, Grindrod KA, Chatterley T, Tsuyuki RT. Paying pharmacists for patient care: A systematic review of remunerated pharmacy clinical care services. Can Pharm J (Ott). 2014 Jul;147(4):209-32. doi: 10.1177/1715163514536678. PMID 25360148
- [Background] Lavikainen P, Aarnio E, Jalkanen K, Tirkkonen H, Rautiainen P, Laatikainen T, Martikainen J. Impact of co-payment level increase of antidiabetic medications on glycaemic control: an interrupted time-series study among Finnish patients with type 2 diabetes. BMC Health Serv Res. 2020 Nov 27;20(1):1095. doi: 10.1186/s12913-020-05952-6. PMID 33246453
- [Background] Houle SK, Grindrod KA, Chatterley T, Tsuyuki RT. Publicly funded remuneration for the administration of injections by pharmacists: An international review. Can Pharm J (Ott). 2013 Nov;146(6):353-64. doi: 10.1177/1715163513506369. PMID 24228051